CLINICAL TRIAL: NCT06783842
Title: Perioperative Depression, an Observational Cohort Study
Status: Active, not recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Max Bell, MD, PhD, Senior Lecturer, Karolinska Institutet
Other Study IDs: 2024-01664-01 Periopdepr
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Surgery With General Anesthesia; Depression - Major Depressive Disorder
Keywords: Perioperative medicine; Perioperative depression; Observational study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgical cohort: Adult patients undergoing surgery

SUMMARY:
This observational cohort study studies two aspects of perioperative depression.

First, it examines the postoperative morbidity and mortality among patients with preoperative depression.

Secondly, in a subset of patients without signs of preoperative depression, the investigators describe the riskfactors for development of de-novo postoperative depression.

DETAILED DESCRIPTION:
BACKGROUND With over 300 million surgeries performed yearly, the impact of perioperative morbidity weighs heavily on society[1]. Multiple studies have highlighted cardiac-[1], renal-[2], pulmonary-[3] and neurological complications[4] as well as other compound metrics of outcome.[5] Postoperative complications, if survived, sometimes result in major impact on function and quality of life.[6] Whilst somatic complications after major surgery are being increasingly investigated, the research field has scarce data on psychological outcomes such as postoperative depression. Most studies use specific surgical cohorts. These include studies of meningioma surgery[7] and glioma patients[8]; both with elevated risk of postoperative depression. In contrast, no significant difference in antidepressant use was found after vestibular schwannoma surgery.[9] When comparing spinal surgery to coronary artery bypass grafting, hysterectomy, cholecystectomy, chronic obstructive pulmonary disease, congestive heart failure exacerbation, and uncomplicated vaginal delivery, the former had the highest risk for postoperative depression.[10] Etiology of major depressive disorder (MDD) is poorly understood, and diagnosis is difficult.[11, 12] Many who experience a first episode of MDD will go on to suffer from recurrent episodes.[13, 14] When compared to equally disabling somatic disorders treatment for depression is less prevalent, indicating under-treatment of the condition.[15] Additionally, individuals with MDD are at elevated risk of cardiovascular disease and all cause-mortality.[16]

HYPOTHESIS The investigators hypothesize that surgery is a stressful event, potentially triggering depression. The investigators further hypothesize that in selected high-risk patients, postoperative new-onset depression is more common and potentially avoidable.

METHODS The investigators plan to use perioperative data from the surgical planning tool, Orbit. The Orbit cohort at Karolinska University Hospital in Solna and in Huddinge, two separate large university hospitals includes Swedish personal identity number (PIN), patient demographics, American Society of Anesthesiologists (ASA) physical status classification, type, date and duration of anesthesia and surgery. NOMESCO classification can be used to subgroup surgical procedures into sixteen categories; neuro, endocrine, ophthalmic, ear, nose and throat, oral and maxillofacial, cardiac, vascular, thoracic, breast, gastrointestinal, urologic, gynecologic, obstetric, orthopedic, dermatologic and minor surgery. The Orbit cohort is cross-matched with electronical medical records (EMR) allowing us to characterize the patients in the cohort based on pre- and postoperative ICD-codes (diagnoses, co-morbid conditions) and pre- and postoperative ATC-codes (medications). Hospital length of stay, readmissions and dates of death can also be retrieved from the EMR.

By merging Orbit data with EMR-data as described above it effectively allows us to investigate short- and long-term outcome for patients developing (new-onset) postoperative depression; this can be achieved by removing patients with depression diagnoses (using ICD-codes from the EMR) and/or patients with collected antidepressants (using ATC-codes from the EMR) in the years prior to surgery. What is the short- and long-term mortality for these patients? How do they far in terms of overall morbidity and health care utilization? The investigators can also characterize the short- and long-term outcome for patients with preoperative depression, focusing specifically on the patients excluded in the study two. How do these patients fare in term of risks for mortality, morbidity and health care utilization?

ELIGIBILITY:
Inclusion Criteria:

*Adult patients (18 years or older) undergoing surgery at Karolinska University Hospital in Solna or in Huddinge

Exclusion Criteria:

*Patients under the age of 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This cohort is fully comprised of adult patients undergoing surgery at Karolinska University Hospital in Solna or in Huddinge
Sampling Method: Probability Sample
Enrollment: 700000 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Mortality | 30/60/90/365-day mortality
  Death after index surgery, time frames (see below)
Days At Home Alive at 30 days after surgery | 30 days
  DAH-30 is calculated using mortality and hospitalisation data from the date of the index surgery (= Day 0). For example, if a patient died on day 2 after their surgery whilst still an inpatient, they would be assigned zero (0) days at home; if a patient was discharged from hospital on Day 6 after surgery but was subsequently re-admitted for 4 days before their second hospital discharge, then they would be assigned a DAH-30 value of 20. If a patient has complications and spends 16 days in hospital, and then is transferred to a nursing facility for rehabilitation, and spend 24 days there before finally being discharged to their own home, they would be assigned a DAH-30 value of zero (0), even though 30-16-24 = -10 because the minimum value of DAH-30 should be zero. If a patient dies within 30 days of surgery, irrespective of whether they have spent some time at home, DAH-30 will be scored as zero (0).
  That is, DAH-30 captures the impact of any complications after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Max Bell, MD, Phd, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data, may be shared to researchers that provide a methodological sound proposal

REFERENCES:
- [Result] Weiser TG, Haynes AB, Molina G, Lipsitz SR, Esquivel MM, Uribe-Leitz T, Fu R, Azad T, Chao TE, Berry WR, Gawande AA. Estimate of the global volume of surgery in 2012: an assessment supporting improved health outcomes. Lancet. 2015 Apr 27;385 Suppl 2:S11. doi: 10.1016/S0140-6736(15)60806-6. Epub 2015 Apr 26. PMID 26313057
- [Result] Prowle JR, Forni LG, Bell M, Chew MS, Edwards M, Grams ME, Grocott MPW, Liu KD, McIlroy D, Murray PT, Ostermann M, Zarbock A, Bagshaw SM, Bartz R, Bell S, Bihorac A, Gan TJ, Hobson CE, Joannidis M, Koyner JL, Levett DZH, Mehta RL, Miller TE, Mythen MG, Nadim MK, Pearse RM, Rimmele T, Ronco C, Shaw AD, Kellum JA. Postoperative acute kidney injury in adult non-cardiac surgery: joint consensus report of the Acute Disease Quality Initiative and PeriOperative Quality Initiative. Nat Rev Nephrol. 2021 Sep;17(9):605-618. doi: 10.1038/s41581-021-00418-2. Epub 2021 May 11. PMID 33976395
- [Result] Fernandez-Bustamante A, Frendl G, Sprung J, Kor DJ, Subramaniam B, Martinez Ruiz R, Lee JW, Henderson WG, Moss A, Mehdiratta N, Colwell MM, Bartels K, Kolodzie K, Giquel J, Vidal Melo MF. Postoperative Pulmonary Complications, Early Mortality, and Hospital Stay Following Noncardiothoracic Surgery: A Multicenter Study by the Perioperative Research Network Investigators. JAMA Surg. 2017 Feb 1;152(2):157-166. doi: 10.1001/jamasurg.2016.4065. PMID 27829093
- [Result] Platzbecker K, Grabitz SD, Raub D, Rudolph MI, Friedrich S, Vinzant N, Kurth T, Weimar C, Bhatt DL, Nozari A, Houle TT, Xu X, Eikermann M. Development and external validation of a prognostic model for ischaemic stroke after surgery. Br J Anaesth. 2021 Nov;127(5):713-721. doi: 10.1016/j.bja.2021.05.035. Epub 2021 Jul 22. PMID 34303492
- [Result] Bell M, Eriksson LI, Svensson T, Hallqvist L, Granath F, Reilly J, Myles PS. Days at Home after Surgery: An Integrated and Efficient Outcome Measure for Clinical Trials and Quality Assurance. EClinicalMedicine. 2019 Apr 27;11:18-26. doi: 10.1016/j.eclinm.2019.04.011. eCollection 2019 May-Jun. PMID 31317130
- [Result] Grocott MP, Pearse RM. Prognostic studies of perioperative risk: robust methodology is needed. Br J Anaesth. 2010 Sep;105(3):243-5. doi: 10.1093/bja/aeq207. No abstract available. PMID 20716567
- [Result] Thurin E, Ryden I, Skoglund T, Smits A, Gulati S, Hesselager G, Bartek J Jr, Henriksson R, Salvesen O, Jakola AS. Impact of meningioma surgery on use of antiepileptic, antidepressant, and sedative drugs: A Swedish nationwide matched cohort study. Cancer Med. 2021 May;10(9):2967-2977. doi: 10.1002/cam4.3868. Epub 2021 Mar 26. PMID 33773085
- [Result] Ryden I, Thurin E, Carstam L, Smits A, Gulati S, Henriksson R, Salvesen O, Store Jakola A. Psychotropic and anti-epileptic drug use, before and after surgery, among patients with low-grade glioma: a nationwide matched cohort study. BMC Cancer. 2021 Mar 8;21(1):248. doi: 10.1186/s12885-021-07939-w. PMID 33685410
- [Result] Thurin E, Forander P, Bartek J Jr, Gulati S, Ryden I, Smits A, Hesselager G, Salvesen O, Jakola AS. Depression and ability to work after vestibular schwannoma surgery: a nationwide registry-based matched cohort study on antidepressants, sedatives, and sick leave. Acta Neurochir (Wien). 2021 Aug;163(8):2225-2235. doi: 10.1007/s00701-021-04862-8. Epub 2021 May 7. PMID 33963435
- [Result] Wilson BR, Tringale KR, Hirshman BR, Zhou T, Umlauf A, Taylor WR, Ciacci JD, Carter BS, Chen CC. Depression After Spinal Surgery: A Comparative Analysis of the California Outcomes Database. Mayo Clin Proc. 2017 Jan;92(1):88-97. doi: 10.1016/j.mayocp.2016.06.030. Epub 2016 Nov 9. PMID 27836112
- [Result] Menard C, Hodes GE, Russo SJ. Pathogenesis of depression: Insights from human and rodent studies. Neuroscience. 2016 May 3;321:138-162. doi: 10.1016/j.neuroscience.2015.05.053. Epub 2015 May 30. PMID 26037806
- [Result] Wancata J, Windhaber J, Bach M, Meise U. Recognition of psychiatric disorders in nonpsychiatric hospital wards. J Psychosom Res. 2000 Feb;48(2):149-55. doi: 10.1016/s0022-3999(99)00098-7. PMID 10719131
- [Result] Eaton WW, Shao H, Nestadt G, Lee HB, Bienvenu OJ, Zandi P. Population-based study of first onset and chronicity in major depressive disorder. Arch Gen Psychiatry. 2008 May;65(5):513-20. doi: 10.1001/archpsyc.65.5.513. PMID 18458203
- [Result] Mueller TI, Leon AC, Keller MB, Solomon DA, Endicott J, Coryell W, Warshaw M, Maser JD. Recurrence after recovery from major depressive disorder during 15 years of observational follow-up. Am J Psychiatry. 1999 Jul;156(7):1000-6. doi: 10.1176/ajp.156.7.1000. PMID 10401442
- [Result] Ormel J, Petukhova M, Chatterji S, Aguilar-Gaxiola S, Alonso J, Angermeyer MC, Bromet EJ, Burger H, Demyttenaere K, de Girolamo G, Haro JM, Hwang I, Karam E, Kawakami N, Lepine JP, Medina-Mora ME, Posada-Villa J, Sampson N, Scott K, Ustun TB, Von Korff M, Williams DR, Zhang M, Kessler RC. Disability and treatment of specific mental and physical disorders across the world. Br J Psychiatry. 2008 May;192(5):368-75. doi: 10.1192/bjp.bp.107.039107. PMID 18450663
- [Result] Rajan S, McKee M, Rangarajan S, Bangdiwala S, Rosengren A, Gupta R, Kutty VR, Wielgosz A, Lear S, AlHabib KF, Co HU, Lopez-Jaramillo P, Avezum A, Seron P, Oguz A, Kruger IM, Diaz R, Nafiza MN, Chifamba J, Yeates K, Kelishadi R, Sharief WM, Szuba A, Khatib R, Rahman O, Iqbal R, Bo H, Yibing Z, Wei L, Yusuf S; Prospective Urban Rural Epidemiology (PURE) Study Investigators. Association of Symptoms of Depression With Cardiovascular Disease and Mortality in Low-, Middle-, and High-Income Countries. JAMA Psychiatry. 2020 Oct 1;77(10):1052-1063. doi: 10.1001/jamapsychiatry.2020.1351. PMID 32520341